CLINICAL TRIAL: NCT05153694
Title: Infectious Complications After Cystectomy: A Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Benedikt Ebner, Resident in Urology, Ludwig-Maximilians - University of Munich
Other Study IDs: RCXINFLMU
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bladder Cancer; Infections; Infection, Bacterial; Infection, Hospital; Infection Wound; Urinary Tract Infections; Urinary Bladder Diseases; Urinary Tract Disease
MeSH Terms: conditions — Urinary Bladder Neoplasms; Infections; Bacterial Infections; Cross Infection; Wound Infection; Urinary Tract Infections; Urinary Bladder Diseases; Urologic Diseases | interventions — Cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cystectomy — Removal of the urinary bladder

SUMMARY:
Patients undergoing cystectomy for either oncological or non-oncological indications are prospectively enrolled following informed consent. This study design incorporates a comprehensive medical history, detailed prospective documentation of clinicopathological parameters, and serial measurements of infectious markers pre- and post-operatively. In-hospital complications are meticulously recorded, and long-term outcomes assessed through structured follow-up interviews at 3, 6, and 12 months. These follow-ups utilize standardized questionnaires to evaluate post-discharge infectious complications and gather patients' perspectives on their in-hospital experiences, providing a robust understanding of both clinical outcomes and patient-reported experiences.

DETAILED DESCRIPTION:
Aims of the study:

1. Prospective evaluation of the association between preoperative interleukin-6 levels and local tumor stage in patients undergoing radical cystectomy
2. Prospective assessment of interleukin-6, procalcitonin and wound drainage culture as early indicators for perioperative infectious complications after cystectomy
3. Prospective evaluation of physician-assessed vs. patient-reported grading of complications after cystectomy
4. Prospective comparison of infectious complications within the first 12 months after cystectomy: ileal neobladder vs. ileal conduit
5. Prospective evaluation of the association between in-hospital complications after cystectomy and quality of life after three months

ELIGIBILITY:
Inclusion Criteria:

* Disease which requires removal of the urinary bladder

Exclusion Criteria:

* Patient does not want to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Infectious parameters on the first postoperative day after cystectomy | First postoperative day
  IL-6 level, procalcitonin level and wound drainage culture
Postoperative fever | Surgery - discharge
  Proportion of cystectomy patients that develops fever postoperatively (≥38.0°C)
Antibiotic use | Surgery - discharge
  Proportion of cystectomy patients that need additional oral or i.v. antibiotic therapy (on top of the hospital standard)
In-hospital complications | Surgery - discharge
  Clavien-Dindo Classification and Comprehensive Complication Index
Antibiotic therapy within the first year after discharge | 0-12 months after discharge
  Proportion of cystectomy patients that needs antibiotic therapy associated with urinary diversion in the first year after discharge
Fever within the first year after discharge | 0-12 months after discharge
  Proportion of cystectomy patients with urinary tract associated fever in the first year after discharge
Emergency consultation | 0-12 months after discharge
  Proportion of cystectomy patients with a cystectomy-associated emergency consultation in the first year after discharge
Inpatient admission | 0-12 months after discharge
  Proportion of cystectomy patients with a cystectomy-associated inpatient admission in the first year after discharge
Preoperative interleukin-6 level | 1 day before surgery
  IL-6 level before surgery

SECONDARY OUTCOMES:
IMCU/ICU nights | Surgery - discharge
  Number of nights spent at a IMCU/ICU postoperatively
Duration of hospital stay | Surgery - discharge
  Total hospital stay (nights)
Subjective grading of in-hospital complications | Assessed time: Surgery - discharge. Assessed 3 months after discharge
  Subjective assessment: no complications, minor complications or major complications
Rating of the pre-operatively provided medical information | Assessed 3 months after discharge
  Subjective assessment: very good, good, satisfactory, sufficient, not sufficient
Health related quality of life | Assessed 3 months after discharge
  EORTC QLQ-C30, FACT-BL- and QLQ-BLM30-questionnaires after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Schulz, PD Dr., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Urology Department - LMU Klinikum, Munich, Outside U.S./Canada, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebner B, Hirsch J, Holz A, Eismann L, Hermans J, Pyrgidis N, Kidess M, Semmler M, Brinkmann I, Aydogdu C, Chaloupka M, Apfelbeck M, Lindner AK, Weinhold P, Stief CG, Volz Y, Schulz GB. Prospective Evaluation of Blood-based and Microbiological Early Indicators of In-hospital Infectious Complications After Open Cystectomy. Eur Urol Open Sci. 2025 Nov 18;83:1-8. doi: 10.1016/j.euros.2025.10.019. eCollection 2026 Jan. PMID 41334533
- [Derived] Ebner B, Hirsch J, Holz A, Volz Y, Eismann L, Hermans J, Pyrgidis N, Kidess M, Semmler M, Fouladgar ST, Papadopoulos I, Chaloupka M, Apfelbeck M, Marcon J, Weinhold P, Ewert A, Kazmierczak P, Stief CG, Schulz GB. Association of interleukin-6 serum levels with local tumor stage and lymph node metastasis of urothelial carcinoma. Urol Oncol. 2025 Dec;43(12):693.e1-693.e8. doi: 10.1016/j.urolonc.2025.08.026. Epub 2025 Sep 25. PMID 41006129
- [Derived] Ebner B, Hirsch J, Holz A, Volz Y, Eismann L, Hermans J, Pyrgidis N, Kidess M, Semmler M, Brinkmann I, Aydogdu C, Chaloupka M, Lindner AK, Weinhold P, Stief CG, Schulz GB. Discrepancies between physician-assessed and patient-reported complications after cystectomy - a prospective analysis. World J Urol. 2025 Feb 10;43(1):115. doi: 10.1007/s00345-025-05487-7. PMID 39928165